CLINICAL TRIAL: NCT01696799
Title: A Multi-Center, Randomized Comparative Study of the Pharmacokinetics of Econazole Nitrate 1% Foam and Econazole Nitrate 1% Cream in Subjects With Interdigital Tinea Pedis Aged 12 Years to Less Than 18 Years
Brief Title: Comparative PK Study of Econazole Nitrate Foam and Econazole Nitrate Cream in Subjects With Interdigital Tinea Pedis Aged 12 Years to Less Than 18 Years
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AmDerma (Industry)
Collaborators: AmDerma Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 079-2951-109
Record Dates: First submitted 2012-09-27; First posted 2012-10-01 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2012-09

CONDITIONS: Interdigital Tinea Pedis
MeSH Terms: interventions — Econazole

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Econazole Nitrate Foam (Experimental): Investigational Drug Product
  Interventions: Drug: Econazole Nitrate
- Vehicle Foam (Placebo Comparator): Vehicle Foam Comparator
  Interventions: Drug: placebo
- Econazole Nitrate Cream (Active Comparator): Active comparator cream product
  Interventions: Drug: Econazole Nitrate

INTERVENTIONS:
Drug: Econazole Nitrate
  Arms: Econazole Nitrate Cream; Econazole Nitrate Foam
Drug: placebo
  Arms: Vehicle Foam

SUMMARY:
To compare the pharmacokinetics of Econazole Nitrate Foam with Econazole Nitrate Cream in subjects with interdigital tinea pedis aged 12 years to less than 18 years.

DETAILED DESCRIPTION:
Based on the results of a previous clinical study evaluating the pharmacokinetics, safety and efficacy of EN Foam versus the reference listed econazole nitrate cream and the foam vehicle in adults, the current clinical study is being conducted to provide additional pharmacokinetic data for EN in the foam formulation in subjects ages 12 to less than 18 years with interdigital tinea pedis to support a clinical bridge for systemic safety to the RLD in this pediatric population. The study also includes clinical and safety endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Be between 12 years and less than 18 years of age and of either sex.
* Have a clinical diagnosis of interdigital tinea pedis
* Parent/guardian has provided written informed consent and the subject has provided written assent.
* Be willing and able to use the assigned study medication as directed and to commit to all follow-up visits for the duration of the study.
* Have microscopic evidence (positive KOH) of the presence of fungi and a positive fungal culture.
* Be in good health and free of any disease or physical condition which might, in the Investigator's opinion, expose the subject to an unacceptable risk by study participation.
* Females must be non-pregnant, non-lactating and not intending to become pregnant during the course of the study.

Exclusion Criteria:

* Is pregnant, nursing or planning a pregnancy during the study
* Has used topical antifungals or topical corticosteroids on the feet within 14 days prior to the start of the study.
* Has received systemic antifungal therapy within 12 weeks prior to the start of the study medication.
* Has used systemic antibacterials or systemic corticosteroids within 14 days prior to the start of the study.
* Has a history of uncontrolled diabetes mellitus or is immunocompromised (due to disease, e.g., HIV, or medications).
* Has concurrent moccasin-type tinea pedis (in the opinion of the Investigator).
* Has any other skin disease which might interfere with the evaluation of tinea pedis.
* Is currently enrolled in an investigational drug or device study.
* Has received an investigational drug or treatment with an investigational device within 30 days prior to entering this study.
* Is unreliable, including subjects with a history of drug or alcohol abuse.
* Has known hypersensitivity to any of the components of the study medications.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2011-09; Primary Completion 2012-04 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Plasma Levels of Econazole Nitrate | 28 Days
  Blood will be taken at Baseline (Day 1) prior to the application of medication, and at the end of treatment (Day 28), just prior to the last dose of medication, and at 7 (±1 hr) hours post-drug application and a third blood draw 4 (±1 hr) hours after the second PK blood draw.
Investigator Assessment of Response to Treatment | 28 Days
  At the end of treatment (Day 28), the Investigator will assess the subject's response to treatment using a 5-point scale (1 = excellent, 2 = very good, 3 = good, 4 = fair, and 5 = poor).

SECONDARY OUTCOMES:
Dosing Compliance | 28 Days
  Measures of study medication compliance will include the total number of applications, duration of treatment, and the total amount of study medication used. The amount of study medication used will be determined post-study following thereturn of all clinical supplies.

CONTACTS AND LOCATIONS:
Locations (1):
- Therapeutics Inc., San Diego, California, United States